CLINICAL TRIAL: NCT00948558
Title: Citrate Pharmacokinetics in Healthy Individuals and Critically Ill Patients and the Application of Regional Citrate Anticoagulation in Continuous Renal Replacement Therapy(RCA-CRRT).
Brief Title: Citrate Pharmacokinetics and Regional Citrate Anticoagulation in CRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Scientific and technology committe (Unknown)
Responsible Party: Feng Ding, Huashan Hospital
Other Study IDs: KY2009-108
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Acute Kidney Failure With or Without:; MODS; Sepsis; Hepatic Insufficiency
Keywords: citrate anticoagulation; pharmacokinetic; critically ill; acute kidney failure
MeSH Terms: conditions — Multiple Organ Failure; Sepsis; Hepatic Insufficiency; Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To compare the differences of citrate pharmacokinetics in healthy individuals and critically ill patients as well as the influential factors.
2. To validate a pharmacokinetic model which has been established in a formal paper.
3. To create a safe and effective RCA-CRRT protocol.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals, none-pregnant
* diagnosed with acute renal failure according to RIFLE criteria
* ARF with hepatic insufficiency
* ARF with MODS or sepsis
* within informed consent

Exclusion Criteria:

* used drugs with citrate within one week
* infused with blood,plasma or platelet or undergone plasma exchange therapy within 48 hours
* serious alkalosis with PH>7.55
* serious lactic acidosis
* not in resuscitation state

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the subjects will be selected from a university teaching hospital in Shanghai, China.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai, China

REFERENCES:
- [Derived] Zheng Y, Xu Z, Zhu Q, Liu J, Qian J, You H, Gu Y, Hao C, Jiao Z, Ding F. Citrate Pharmacokinetics in Critically Ill Patients with Acute Kidney Injury. PLoS One. 2013 Jun 18;8(6):e65992. doi: 10.1371/journal.pone.0065992. Print 2013. PMID 23824037